CLINICAL TRIAL: NCT00870350
Title: An Immunogenicity and Safety Study of Combined Adsorbed Tetanus, Low Dose Diphtheria and Acellular Pertussis Vaccine (Td5ap and Td1aP) Given as a School-leaving Booster to 14-15-year-old Children Primed With a Five Component Acellular Pertussis Vaccine at 3, 5 and 12 Months of Age, and a Booster Dose at 5½ Years of Age
Brief Title: An Immunogenicity and Safety Study of Tetanus, Diphtheria and Acellular Pertussis Vaccine Booster
Acronym: Tdap Booster
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swedish Institute for Infectious Disease Control (Other)
Collaborators: MCM Vaccines B.V. (Industry); Statens Serum Institut (Other)
Responsible Party: Prof. em. Leif Gothefors, Swedish Institute for Infectious Disease Control
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-008195-13
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2009-03

CONDITIONS: Tetanus; Diphtheria; Pertussis
Keywords: immunogenicity; safety; tetanus; diphtheria; acellular; pertussis; vaccine; booster; adverse event; adverse reaction; DT1aP; DT5ap; FHA; fimbriae; pertactin; SMI; Smittskyddsinstitutet; Immune response and safety profile to a Tdap booster
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Td5ap (Active Comparator): Group 1 receiving Td5ap as a single intramuscular injection.
  Interventions: Biological: Td5ap
- Td1aP (Active Comparator): Group 2 receiving Td1aP as a single intramuscular injection
  Interventions: Biological: Td1aP

INTERVENTIONS:
Biological: Td5ap — Intramuscular injection of 0.5 mL Td5ap (COVAXiS) on day 1.
  Other Names: COVAXiS
  Arms: Td5ap
Biological: Td1aP — Intramuscular injection of 0.5 mL Td1aP (diTekiBooster) on day 1.
  Other Names: diTekiBooster
  Arms: Td1aP

SUMMARY:
Open-label, randomized, multi-centre study in which 400 subjects, divided into two groups, will receive Td5ap or Td1aP as a single injection. We will then describe the immune response and safety profile of the combined vaccine booster.

DETAILED DESCRIPTION:
The vaccines in the study are COVAXIS (Td5ap), Sanofi Pasteur Canada, and diTekiBooster (Td1aP), Statens Serum Institut, Denmark.

The primary objective of the study is to describe the immune response to diphtheria toxin, tetanus toxoid, pertussis toxin, filamentous haemagglutinin (FHA), fimbriae 2/3 and pertactin four weeks after immunization with Td1aP and Td5ap.

The secondary objectives include:

* describing the safety of a fith dose of DTP vaccines in 14-15 year-old children by observing systemic and local adverse reactions
* describing pre-booster antibody levels
* describing pre-booster and post-booster IgG and IgA levels in saliva
* describing in a subpopulation the pre-booster and post-booster T cell immune responses as determined by the production of cytokines
* describing in a subpopulation the pre-booster and post-booster B cell immune responses as determined by the number of effector and memory B-cells

The sample size is 400 subjects (200 in group 1 and 200 in group 2). It will be an open-label, randomized, multi-centre study in which group 1 will receive Td5ap as a single injection and group 2 will receive Td1aP as a single injection. DTP antibodies will be measured before and 28 days (+ 14 days) after Td5ap and Td1aP vaccination. The proportion of children with positive IgG antibody response will be measured in each study arm. Sera will be tested blindly by established ELISA methods and saliva samples will be analyzed by exploratory assays. In a subpopulation cellmediated immunity will be analyzed. The safety evaluation criteria will be the percentage of subjects with adverse events describing injection-site adverse reactions, systemic adverse events, daily temperatures and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject
* 14-15 years old
* eligible for their school-leaving booster for DTP
* received a complete primary vaccination with a 5-component acellular pertussis vaccine (DT5aP-IPV-Hib) at 3, 5 and 12 months of age and vaccinated with a 5-component acellular pertussis vaccine (Td5aP-IPV or Td5aP + IPV) as a booster at 5½ years of age
* informed consent form signed by the subject and parent(s)/legal representative
* subject understand and comply with the study procedures (i.e. able to read and write Swedish)
* female must provide an agreement that they are either sexually continent or practice adequate contraceptive methods (intra-uterine contraceptive device (IUCD), hormonal contraceptives, condoms or other adequate barrier contraception).

Exclusion Criteria:

* acute febrile illness or axillary temperature ≥38.0°C at the time of vaccination
* receipt of immunoglobulin within the previous 3 months, immunosuppression (e g evidence of impaired cell mediated immunity, receipt of immunosuppressant drugs within the previous 3 months or receipt of systemic corticosteroids given daily or on alternate days at ≥20 mg/day prednisone equivalent during >14 days within the past 30 days)
* receipt of a non-study vaccine in the past 30 days
* evolving encephalopathy not attributable to another identifiable cause within 7 days of administration of a previous dose of any vaccine
* booster vaccination with tetanus, low dose diphtheria and acellular pertussis vaccine since the booster vaccination at 5½ years of age
* previous clinical or bacteriological diagnosis of diphtheria, tetanus or pertussis
* hypersensitivity to any component of any of the study vaccines
* current participation in any other clinical trial or participation in any clinical trial in the previous month
* inability to adhere to the protocol, including plans to move from the area
* severe chronic disease
* family history of congenital or hereditary immunodeficiency
* any sever thrombocytopenia or any other coagulation disorder that would contraindicate intramuscular injection
* any medical condition, which in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
to describe in each arm the immune response to diptheria toxin, tetanus toxoid, pertussis toxin, FHA, fimbriae 2/3 and pertactin four weeks after immunization with Td1aP and Td5ap | 42 days

SECONDARY OUTCOMES:
safety of a fith dose of DTP vaccines | 42 days
pre-booster antibody levels | 42 days
pre-booster and post-booster IgG and IgA levels | 42 days
pre-booster and post-booster T cell immune responses | 42 days
pre-booster and post-booster B cell immune responses | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Leif Gothefors, Prof. em., Principal Investigator — Swedish Institute for Infectious Disease Control; Eva Netterlid, Study Director — Swedish Institute for Infectious Disease Control
Locations (1):
- Swedish Institute for Infectious Disease Control, Lund, Sweden

REFERENCES:
- [Derived] Lin A, Apostolovic D, Jahnmatz M, Liang F, Ols S, Tecleab T, Wu C, van Hage M, Solovay K, Rubin K, Locht C, Thorstensson R, Thalen M, Lore K. Live attenuated pertussis vaccine BPZE1 induces a broad antibody response in humans. J Clin Invest. 2020 May 1;130(5):2332-2346. doi: 10.1172/JCI135020. PMID 31945015
- [Derived] Carlsson RM, Gustafsson L, Hallander HO, Ljungman M, Olin P, Gothefors L, Nilsson L, Netterlid E. Two consecutive randomized controlled pertussis booster trials in children initially vaccinated in infancy with an acellular vaccine: The first with a five-component Tdap vaccine to 5-year olds and the second with five- or monocomponent Tdap vaccines at age 14-15 years. Vaccine. 2015 Jul 17;33(31):3717-25. doi: 10.1016/j.vaccine.2015.05.079. Epub 2015 Jun 7. PMID 26057135
- [Derived] Jahnmatz M, Ljungman M, Netterlid E, Jenmalm MC, Nilsson L, Thorstensson R. Pertussis-specific memory B-cell and humoral IgG responses in adolescents after a fifth consecutive dose of acellular pertussis vaccine. Clin Vaccine Immunol. 2014 Sep;21(9):1301-8. doi: 10.1128/CVI.00280-14. Epub 2014 Jul 9. PMID 25008903